CLINICAL TRIAL: NCT02200146
Title: Hydroxychloroquine as Steroid-Sparing Agent in Pulmonary Sarcoidosis (HySSAS). A Multicenter, Prospective, Controlled, Randomized Trial.
Brief Title: Hydroxychloroquine as Steroid-Sparing Agent in Pulmonary Sarcoidosis (HySSAS).
Acronym: HySSAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HySSAS-FARM639KLZ
Record Dates: First submitted 2014-07-10; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Sarcoidosis
Keywords: sarcoidosis; treatment; lung; glucocorticoids; hydroxychloroquine
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Prednisone; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Active Comparator): Prednisone per os 0,5 mg/kg/die once/day for 3 months. After 3 months, between responders, prednisone was slowly tapered (5 mg/week maintaining the new reduced dose for one week) to 0,2 mg/kg/die for further 6 months.
  Interventions: Drug: Prednisone
- Hydroxychloroquine + Prednisone (Experimental): Hydroxychloroquine per os 200 mg/die (or adjusted for body weight if less than 61 kg), twice/day + prednisone 0,15 mg/kg per os daily, once/day for 3 months, than for further 6 months between responders.
  Interventions: Drug: Hydroxychloroquine + Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone per os 0,5 mg/kg/die once/day for 3 months. After 3 months, between responders, prednisone was slowly tapered (5 mg/week maintaining the new reduced dose for one week) to 0,2 mg/kg/die for further 6 months.
  Arms: Prednisone
Drug: Hydroxychloroquine + Prednisone — Hydroxychloroquine per os 200 mg/die (or adjusted for body weight if less than 61 kg), twice/day + prednisone 0,15 mg/kg per os daily, once/day for 3 months, than for further 6 months between responders.
  Arms: Hydroxychloroquine + Prednisone

SUMMARY:
The aim of the study is determining the non-inferiority in the overall success rate and the safety for a combination therapy with hydroxychloroquine plus low dose glucocorticoids compared to that for high dose glucocorticoids at 3 and 9 months in patients with pulmonary sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 70 years
* parenchymal pulmonary involvement at Chest X-Ray (CXR) AND one of the follows: physiologic abnormalities on pulmonary function testing and/or respiratory symptoms, and/or exercise-induced abnormalities.

Exclusion Criteria:

* Unable to understand protocol and to sign informed consent or not suitable candidate to comply with the requirements of this study, in the opinion of the investigator
* Cardiac and neurological sarcoidosis or any other organ involvement
* End stage lung disease at high-resolution computed tomography (HRCT)
* Clinical evidence of active infection
* Documented exposure to beryllium
* Patients with Forced Expiratory Volume at one second (FEV1) changes after salbutamol inhalation ≥20%
* Comorbidity: advanced liver cirrhosis or abnormal liver function, unstable cardiac disease, moderate to severe renal insufficiency, poorly controlled diabetes
* Pregnancy or lactation
* A tuberculin skin test (5 I.U.) more than 5 mm
* Psoriasis
* Homozygous glucose-6-phosphatase deficiency
* Known hypersensitivity to hydroxychloroquine or 4-aminoquinoline derivatives
* Visual field changes attributable to 4-aminoquinolines
* Concomitant therapies: any patient enrolled in the study must be off all prohibited medications at least 4 weeks before screening. Once patients completed the washout period, they may enter the screening period that may last up to 30 days
* Previous therapies: any patient enrolled must be off all medications for sarcoidosis at least 4 weeks before screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-03; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The primary EFFICACY measure is the per-subject overall success rate at the 3 month visit. Overall response is defined as a combined radiographic and clinical responses. | Baseline- After 3 months of treatment
  Subjects is considered clinically cured at the 3 month visit if they will have radiographic success (determined if Chest X-Ray is resolved or improved compared to the baseline; improvement was assessed if there were reduction in hilar adenopathies, less pulmonary involvement, changing in radiographic stage) PLUS a change in at least one of the followings: symptoms (determined by dyspnea or cough index score decrease compared to the baseline), and/or functional improvement (determined by an increase in % of predicted Forced Vital Capacity and/or increase in % of predicted Single-Breath Diffusion capacity of Lung for Carbon monoxide DLCO-SB compared to the baseline), and/or increase in resting Partial pressure of Oxygen in the artery blood (PaO2), and/or worst oxygen saturation increase during 6 Minute Walk Test (6MWT) and/or increase in distance walked at 6MWT, compared to the baseline
The primary SAFETY endpoint is the percent change in lumbar spine (L1-L4) bone mineral density from baseline to month 9 as measured by Dual energy X-ray Absorptiometry (DXA) | Baseline - After 9 months of treatment

SECONDARY OUTCOMES:
Secondary EFFICACY endpoint was the change from baseline in radiographic success rate after 9 month of therapy (measured by High Resolution Chest Tomography HRCT) | Baseline- After 9 months of therapy
  The radiographic success is determined if HRCT is resolved or improved compared to the baseline after 9 months
Secondary SAFETY endpoint was the change from baseline in Body Mass Index | Baseline - After 3, 6 and 9 months
Secondary SAFETY endpoint was the change from baseline in HbA1c | At 3, 6 and 9 months of therapy
Secondary SAFETY endpoint was the change from baseline in clinical laboratory tests (including inflammatory markers) | At 3, 6 and 9 months of therapy
Secondary SAFETY endpoint was the change from baseline in bone turnover markers and mineral metabolism | At months 3 and 9 from the start of therapy
Secondary safety endpoint was the number of participants with Serious and Non-Serious Adverse Events | Within the 9 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pesci, Principal Investigator — Università Milano Bicocca
Locations (1):
- Università degli Studi di Milano - Bicocca, Milan, Milano, Italy